CLINICAL TRIAL: NCT01643382
Title: Randomized Study of the Impact of Peri-operative Glucose Control on Short Term Renal Allograft Function After Transplantation
Brief Title: Hyperglycemia in Renal Transplantation
Acronym: HiRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HiRT 042918
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Diabetes; End Stage Renal Disease
Keywords: diabetes; kidney transplant; end stage renal disease; delayed draft function
MeSH Terms: conditions — Diabetes Mellitus; Kidney Failure, Chronic | interventions — Insulin; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tight glucose control (Experimental): Patients randomized to the tight glucose control arm will be placed on an insulin infusion, or continuous low dose insulin drip.
  Interventions: Drug: Insulin
- Standard glucose control (Active Comparator): Patients randomized to the standard glucose control group will be given subcutaneous doses of insulin every few hours based on their blood sugar.
  Interventions: Drug: Insulin, Asp(B28)-

INTERVENTIONS:
Drug: Insulin — Insulin will be given in a continuous low dose infusion. The infusion will be adjusted based on the patient's blood sugar with the goal of keeping the level between 100-140 mg/dL
  Arms: Tight glucose control
Drug: Insulin, Asp(B28)- — Insulin will be given through subcutaneous injection every few hours based on the patient's blood sugar level.
  Arms: Standard glucose control

SUMMARY:
Based on multiple prior studies, kidney transplant recipients with diabetes are at higher risk for poor initial graft function after transplant. Our study is designed to determine if tight blood sugar control around the time of kidney transplant will improve short term graft function.

DETAILED DESCRIPTION:
Population- Our study population will include all adult diabetic patients undergoing deceased donor renal transplantation or living donor transplantation in which a swap requires transportation and resulting cold storage time. This will ensure a reasonable incidence of our primary outcome (poor short term graft function) and eliminate the potential risk of treating non-diabetic patients with insulin infusions. Patients already enrolled in a drug trial designed to study the impact of the drug on graft function will be excluded.

Study Design- This will be a randomized control trial. Recipients will be randomized to either tight peri-operative glucose control or standard management.

Methods

Randomization Protocol- In order to ensure that patients are equally distributed between groups, we will use block randomization. Blocks of 4 patients will be created with the total number of experimental versus control assignments being equal across blocks. Patients will then be randomly assigned to a block.

Interventions- The study group will be treated with an insulin infusion to achieve tight glycemic control (100-140mg/dL). Each study patient will be started on an insulin infusion prior to their operation. This infusion will continue throughout the operation and for 24 hours after completion of the transplant. Glucose control will then be left to the discretion of the primary team.

The control group will be treated with bolus insulin based on a standard insulin sliding scale.

Outcomes

Aim 1-

Primary endpoint- Our primary endpoint will be poor initial graft function defined by the occurrence of DGF (defined by a decrease in serum creatinine of <10%/day for 3 consecutive days after transplant) or slow graft function (serum creatinine >3 mg/dL 5 days after transplant without dialysis)

Secondary endpoint- Secondary endpoints will include wound infection, length of hospital stay, 30 day mortality, hypoglycemic episodes(glucose <70 mg/dL) and stroke.

Aim 2-

Primary endpoint- Our primary endpoints will be acute rejection at 90 days and graft survival/renal function at 3months, 6months and then yearly.

Statistical Analysis- Data will be described as means with standard deviations or percentages with ranges based on whether the data represent continuous or categorical variables. The t-test and chi-squared test will be used to test hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* diabetic
* end stage renal disease undergoing cadaveric renal transplant

Exclusion Criteria:

* enrolled in concurrent study to test impact of a drug on graft function after transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Parekh, MD, MAS, Principal Investigator — UCSF Department of Surgery
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Parekh J, Niemann CU, Dang K, Hirose R. Intraoperative hyperglycemia augments ischemia reperfusion injury in renal transplantation: a prospective study. J Transplant. 2011;2011:652458. doi: 10.1155/2011/652458. Epub 2011 Sep 4. PMID 21904663
- [Background] Parekh J, Bostrom A, Feng S. Diabetes mellitus: a risk factor for delayed graft function after deceased donor kidney transplantation. Am J Transplant. 2010 Feb;10(2):298-303. doi: 10.1111/j.1600-6143.2009.02936.x. Epub 2010 Jan 6. PMID 20055796
- [Result] Parekh J, Roll GR, Wisel S, Rushakoff RJ, Hirose R. Effect of moderately intense perioperative glucose control on renal allograft function: a pilot randomized controlled trial in renal transplantation. Clin Transplant. 2016 Oct;30(10):1242-1249. doi: 10.1111/ctr.12811. Epub 2016 Sep 24. PMID 27423055
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tight Glucose Control | Standard Glucose Control
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tight Glucose Control | Standard Glucose Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.1) | 60.7 (11) | 60.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 20 | 20 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 5 | 7
  Hispanic | 11 | 13 | 24
  Black | 3 | 6 | 9
  Asian/Islander | 13 | 6 | 19
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Duration dialysis [Mean (Standard Deviation); unit: years] | 5.9 (2.6) | 5.7 (2.7) | 5.8 (3.7)
Duration diabetes [Mean (Standard Deviation); unit: years] | 18.6 (11) | 21.1 (9.9) | 19.9 (14.2)
Hemoglobin A1C [Mean (Standard Deviation); unit: percent hemoglobin] | 6.5 (1.2) | 6.7 (1) | 6.6 (1.6)
Preoperative diabetic regimen [Count of Participants; unit: Participants]
  Insulin | 17 | 17 | 34
  Oral | 6 | 7 | 13
  None | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Poor Graft Function After Kidney Transplant
Description: Our primary endpoint will be poor initial graft function defined by the occurrence of DGF (defined by a decrease in serum creatinine of <10%/day for 3 consecutive days after transplant) or slow graft function (serum creatinine >3 mg/dL 5 days after transplant without dialysis)
Time Frame: 7 days after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Tight Glucose Control | Standard Glucose Control
Number analyzed (Participants) | 30 | 30
Participants | 13 | 22

ADVERSE EVENTS:
Arm/Group | Tight Glucose Control | Standard Glucose Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 2/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes